CLINICAL TRIAL: NCT02651909
Title: Utilization of Thromboelastography to Monitor Rivaroxaban Activity in Trauma and Emergency Surgery Patients
Brief Title: Utilization of TEG to Monitor Rivaroxaban Activity
Status: Completed | Type: Observational
Sponsor: Matthew Neal MD (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, Matthew Neal MD, Matthew D. Neal, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: PRO15050224
Record Dates: First submitted 2015-06-15; First posted 2016-01-11 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Anemia; Venous Thrombosis
MeSH Terms: conditions — Anemia; Venous Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rivaroxaban Cohort: Evidence of Rivaroxaban use with-in the last 48hours Participating subjects will not undergo any procedures associated with this study except data collection and minimal blood sampling of which results will not be become part of the medical record and no clinical decisions will be made using the results of research lab results. Blood samples are for TEG analysis and for Thrombin time, thrombin generation, PT with neoplastine, ecarin chromogenic assay, anti-factor Xa (rivaroxaban assay
  Interventions: Other: blood sampling
- Control cohort not taking Rivaroxaban: Not taking Rivaroxaban - matched to Rivaroxaban group by age gender, type of injury or illness requiring urgent surgery Participating subjects will not undergo any procedures associated with this study except data collection and minimal blood sampling of which results will not be become part of the medical record and no clinical decisions will be made using the results of research lab results. Blood samples are for TEG analysis and for Thrombin time, thrombin generation, PT with neoplastine, ecarin chromogenic assay, anti-factor Xa (rivaroxaban assay
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — blood sampling for TEG analysis, Thrombin time, thrombin generation, PT with neoplastine, ecarin chromogenic assay, anti-factor Xa (rivaroxaban assay

SUMMARY:
The invesigators seek to devise a strategy for the assessment of Rivaroxaban activity in trauma and Emergency General Surgery (EGS) patients available as point-of-care testing.

Thromboelastography (TEG) is a point of care, viscoelastic measurement of coagulation that is widely used in trauma and is viewed by many as superior to standard coagulation studies for the assessment of coagulopathy following injury and may be useful in detecting rivaroxaban effect in trauma and EGS patients to assess the degree of functional factor Xa impairment.

DETAILED DESCRIPTION:
Rivaroxaban is a novel factor Xa inhibitor that is widely used for stroke prevention in nonvalvular atrial fibrillation, treatment of venous thromboembolism (VTE), and for VTE prophylaxis in patients undergoing knee or hip replacement surgery.

Current standard measurements of coagulation are relatively poor at reliably measuring detecting Rivaroxaban effects and more elaborate means of testing such as measurement of factor Xa activity are not immediately available so not useful in Urgent situations such as traumatic injury or emergent surgical indications. Due to the unmet need to devise a strategy for detecting Rivaroxaban activity in urgent situations, unnecessary reversal, which can lead to significant complications and cost, often results.

The investigators seek to devise a strategy for the assessment of Rivaroxaban activity in trauma and Emergency General Surgery (EGS) patient available as point-of-care testing.

Thromboelastography (TEG) is a point of care, viscoelastic measurement of coagulation that is widely used in trauma and is viewed by many as superior to standard coagulation studies for the assessment of coagulopathy following injury and may be useful in detecting Rivaroxaban effect in trauma and EGS patients to assess the degree of functional factor Xa impairment.

This proposed study is a observational, prospective, cross sectional, study evaluating the Pharmacokinetics of rivaroxaban utilization thromboelastography (TEG) in a population of 80 trauma and emergency EGS patients who were taking rivaroxaban prior to admission and 20 active control trauma and EGS patients who were not taking rivaroxaban prior to admission (matched by age gender injury mechanism or illness)

Study activities:

Prior to any resuscitation with blood, blood products, or reversal agents, the investigators will obtain a TEG as well as standard coagulation testing: prothrombin time, partial thromboplastin time,international normalized ratio (PT/PTT/INR). TEG and coagulation studies will be obtained as soon as possible on admission and again following reversal of rivaroxaban (if reversed as SOC) or at 24 hours post admission to assess for changes.

To assess the efficacy of TEG in monitoring Rivaroxaban activity, the investigators will also perform a battery of coagulation tests at the same timepoints described above in order to attempt to assess the degree of functional factor X inhibition. The coagulation battery will include: thrombin time, thrombin generation, PT with neoplastine, ecarin chromogenic assay, as well as the anti-factor Xa chromogenic assay (Rivaroxaban assay) run by our Institute for Transfusion Medicine.

TEG will be compared to these additional coagulation assays to determine whether prolongation of R time (the most sensitive measurement of coagulation factor activity) and other TEG parameters can be utilized as reliable measurements of Rivaroxaban activity. Each of these tests will be performed at the two aforementioned timepoints: admission and post reversal or 24 hours post admission if clinical team does not opt to reverse patent.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Evidence of Rivaroxaban use with-in the last 48hours per medical records or report by patient, family, or other healthcare member familiar with patients drug medical history
3. Willingness of subject or legally authorized representative to provide written consent for study procedures.

Exclusion Criteria:

1. Known to be pregnant
2. Known to be a prisoner
3. Known Chronic liver disease
4. Documented hypo coagulation condition (hemophilia, Von Willebrands, any congenital factor deficiency (V,X,XII) leukemia)
5. Use of any anticoagulant medication other than Rivaroxaban (examples: Warfarin, lovenox, arixtra, fragmin, eliquis)
6. Prehospital blood product administration (FFP, platelets, Prothrombin Complex Concentrate (PCC), tranexamic acid (TXA)
7. Non-survivable traumatic brain Injury
8. Comfort Measure Only (CMO) status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have taken the drug Rivaroxaban with-in the past 48hours that arrive in the ED with traumatic injury or with illness requiring emergent surgery
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-04; Primary Completion 2018-07-07 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Change in thromboelastography (TEG) as a measure of anticoagulation following Rivaroxaban reversal in trauma and emergency general surgery patients | 2 time-points: First TEG immediately upon presentation to the emergency department - 2nd timepoint is within 1 hour of Rivaroxaban reversal
  To best observe inhibition of factor Xa, the investigators will perform kaolin TEGs as opposed to alternative forms of activated TEG (rapid-TEG) which may artificially induce coagulation and miss an effect on factor Xa activity. Additional TEG formats that may better target factor Xa inhibition will be investigated in parallel. As a control group, a second cohort of trauma and EGS patients (matched by demographics, injury mechanism, and illness) who are not taking Rivaroxaban will be identified. TEG and coagulation studies will be obtained on admission as described above. Following reversal of Rivaroxaban for subjects that a clinical decision is made to give reversal agents, or at 24 hours post admission for all other subjects, the TEG and PT/PTT/INR will be repeated to assess for changes in both groups.

SECONDARY OUTCOMES:
TEG as a point-of-care analysis following Rivaroxaban as compared to the standard of care measurement of coagulation. | 2 time-points: First TEG immediately upon presentation to the emergency department - 2nd timepoint is within 1 hour of Rivaroxaban reversal
  To assess the efficacy of TEG in monitoring Rivaroxaban activity, the investigators will perform a battery of coagulation tests in order to attempt to assess the degree of functional factor X inhibition. The coagulation battery will include: thrombin time, thrombin generation, PT with neoplastine, INR, PTT, ecarin chromogenic assay, as well as the anti-factor Xa chromogenic assay (Rivaroxaban assay) run by the Institute for Transfusion Medicine at the University of Pittsburgh. TEG will be compared to these additional coagulation assays to determine whether prolongation of R time (the most sensitive measurement of coagulation factor activity) and other TEG parameters can be utilized as reliable measurements of Rivaroxaban activity. Each of these tests will be performed at the two aforementioned time points: admission and post-reversal/24 hours post admission

OTHER OUTCOMES:
Clinical Outcomes data to be collected from Subject's medical records | During entire duration of hospital stay, an expected average of 30 days:
  1. Bleeding complications
  2. Transfusion requirements (red blood cells and blood components)
  3. Use, effects and costs of reversal agents
  4. Use of tranexamic acid
  5. Surgical or interventional procedures performed with outcome
  6. Incidence of venous thromboembolism (VTE)
  7. Management and timing of VTE prophylaxis
  8. Nosocomial infections
  9. Mortality
  10. ICU and hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Neal, MD, Principal Investigator — University of Pittsburgh, Division of Trauma and Acute Care Surgery Department of Surgery
Locations (1):
- University of Pittsburgh Medical Center, PUH, 200 Lothrop Street, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Piccini JP, Hellkamp AS, Lokhnygina Y, Patel MR, Harrell FE, Singer DE, Becker RC, Breithardt G, Halperin JL, Hankey GJ, Berkowitz SD, Nessel CC, Mahaffey KW, Fox KA, Califf RM; ROCKET AF Investigators. Relationship between time in therapeutic range and comparative treatment effect of rivaroxaban and warfarin: results from the ROCKET AF trial. J Am Heart Assoc. 2014 Apr 22;3(2):e000521. doi: 10.1161/JAHA.113.000521. PMID 24755148
- [Background] Beyer-Westendorf J, Lutzner J, Donath L, Tittl L, Knoth H, Radke OC, Kuhlisch E, Stange T, Hartmann A, Gunther KP, Weiss N, Werth S. Efficacy and safety of thromboprophylaxis with low-molecular-weight heparin or rivaroxaban in hip and knee replacement surgery: findings from the ORTHO-TEP registry. Thromb Haemost. 2013 Jan;109(1):154-63. doi: 10.1160/TH12-07-0510. Epub 2012 Nov 29. PMID 23197272
- [Background] Gordon JL, Fabian TC, Lee MD, Dugdale M. Anticoagulant and antiplatelet medications encountered in emergency surgery patients: a review of reversal strategies. J Trauma Acute Care Surg. 2013 Sep;75(3):475-86. doi: 10.1097/TA.0b013e3182a07391. No abstract available. PMID 24089118
- [Background] Holcomb JB, Minei KM, Scerbo ML, Radwan ZA, Wade CE, Kozar RA, Gill BS, Albarado R, McNutt MK, Khan S, Adams PR, McCarthy JJ, Cotton BA. Admission rapid thrombelastography can replace conventional coagulation tests in the emergency department: experience with 1974 consecutive trauma patients. Ann Surg. 2012 Sep;256(3):476-86. doi: 10.1097/SLA.0b013e3182658180. PMID 22868371
- [Background] Muller MC, Meijers JC, Vroom MB, Juffermans NP. Utility of thromboelastography and/or thromboelastometry in adults with sepsis: a systematic review. Crit Care. 2014 Feb 10;18(1):R30. doi: 10.1186/cc13721. PMID 24512650
- [Background] Bowry R, Fraser S, Archeval-Lao JM, Parker SA, Cai C, Rahbar MH, Grotta JC. Thrombelastography detects the anticoagulant effect of rivaroxaban in patients with stroke. Stroke. 2014 Mar;45(3):880-3. doi: 10.1161/STROKEAHA.113.004016. Epub 2014 Jan 14. PMID 24425115